CLINICAL TRIAL: NCT02027337
Title: The Changes of Hemocoagulation and Lipoperoxidation in Women Using Combined Oral Contraceptives With Antiandrogenic Activity, Correction by Antioxidants
Brief Title: Hemocoagulation and Lipoperoxidation in Women Using Combined Oral Contraceptives, Correction by Antioxidants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tyumen State Medical Academy (Other)
Responsible Party: Principal Investigator, Khvoschina Tatyana N., Tyumen State Medical Academy, Tyumen State Medical Academy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01200707998
Record Dates: First submitted 2013-12-26; First posted 2014-01-06 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-01

CONDITIONS: Polycystic Ovarian Syndrome; Hyperandrogenism; Menstrual Irregularities
Keywords: combined oral contraceptives; drospirenone; cyproterone; hemostasis; antioxidants
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism; Menstruation Disturbances | interventions — Ethinyl Estradiol; drospirenone and ethinyl estradiol combination; Cyproterone acetate, ethinyl estradiol drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Control group (No Intervention): Healthy women that no use combined oral contraceptives
- 20 mcg EE/3 mg drospirenone (Experimental): Women that use combined oral contraceptives containing 20 mcg ethinylestradiol/3 mg drospirenone (Yaz)
  Interventions: Drug: 20 mcg ethinylestradiol /3 mg drospirenone
- 20 mcg EE/3 mg drospirenone and Selmevit (Experimental): Women that use combined oral contraceptives containing 20 mcg ethinylestradiol/3 mg drospirenone (Yaz) and antioxidant complex Selmevit
  Interventions: Drug: 20 mcg ethinylestradiol/3 mg drospirenone and Selmevit
- 30 mcg EE/3 mg drospirenone (Experimental): Women that use combined oral contraceptives containing 30 mcg ethinylestradiol/3 mg drospirenone (Yasmin)
  Interventions: Drug: 30 mcg ethinylestradiol/3 mg drospirenone
- 30 mcg EE/3 mg drospirenone and Selmevit (Experimental): Women that use combined oral contraceptives containing 30 mcg ethinylestradiol/3 mg drospirenone (Yasmin) and antioxidant complex Selmevit
  Interventions: Drug: 30 mcg ethinylestradiol/3 mg drospirenone and Selmevit
- 35 mcg EE/2mg cyproterone (Experimental): Women that use combined oral contraceptives containing 35 mcg ethinylestradiol/2 mg cyproterone
  Interventions: Drug: 35 mcg ethinylestradiol/2 mg cyproterone
- 35 mcg EE/2 mg cyproterone and Selmevit (Experimental): Women that use combined oral contraceptives containing 20 mcg ethinylestradiol/2 mg cyproterone and Selmevit
  Interventions: Drug: 35 mcg ethinylestradiol/2 mg cyproterone and Selmevit

INTERVENTIONS:
Drug: 20 mcg ethinylestradiol /3 mg drospirenone — One contraceptive pill in each day of 28 day cycle. Number of Cycles: 12
  Other Names: Yaz
  Arms: 20 mcg EE/3 mg drospirenone
Drug: 20 mcg ethinylestradiol/3 mg drospirenone and Selmevit — One contraceptive pill in each day of 28 day cycle. Number of Cycles: 12. Two pills of Selmevit in each day during 30 days, repeat of the course every 3 months.
  Other Names: Yaz; Selmevit
  Arms: 20 mcg EE/3 mg drospirenone and Selmevit
Drug: 30 mcg ethinylestradiol/3 mg drospirenone — One contraceptive pill in each of 21 days, than 7 days break. Number of Cycles: 12
  Other Names: Yasmin
  Arms: 30 mcg EE/3 mg drospirenone
Drug: 30 mcg ethinylestradiol/3 mg drospirenone and Selmevit — One contraceptive pill in each of 21 days, than 7 days break. Number of Cycles: 12 Two pills of Selmevit in each day during 30 days, repeat of the course every 3 months.
  Other Names: Yasmin; Selmevit
  Arms: 30 mcg EE/3 mg drospirenone and Selmevit
Drug: 35 mcg ethinylestradiol/2 mg cyproterone — 1 contraceptive pill in each day of 28 day cycle. Number of Cycles: 12
  Other Names: Diane-35; Chloe
  Arms: 35 mcg EE/2mg cyproterone
Drug: 35 mcg ethinylestradiol/2 mg cyproterone and Selmevit — One contraceptive pill in each day of 28 day cycle. Number of Cycles: 12. Two pills of Selmevit in each day during 30 days, repeat of the course every 3 months.
  Other Names: Diane-35; Chloe; Selmevit
  Arms: 35 mcg EE/2 mg cyproterone and Selmevit

SUMMARY:
We investigate parameters of hemocoagulation and lipoperoxidation in women using combined oral contraceptives with antiandrogenic activity (containing drospirenone with 20 or 30 mcg ethinylestradiol; or cyproterone acetate); correction of these changes by antioxidants

DETAILED DESCRIPTION:
It is well known that hormonal contraceptives using increase risk of thrombosis. We conduct parameters of hemostasis in women that use combined oral contraceptives with antiandrogenic activity for contraception and treatment. Considering relationship between lipoperoxidation in platelets and hemostasis we expect that limitation of lipoperoxidation by antioxidants can restrict hypercoagulation and decrease risk of thrombosis.

The purpose of this study is decrease of thrombosis risk in women that use combined oral contraceptives containing 20 mcg ethinylestradiol/3 mg drospirenone, 30 mcg ethinylestradiol/3 mg drospirenone, 35 mcg ethinylestradiol/2mg cyproterone acetate. Half of the women of each arm (group) receive only combined oral contraceptives (COC), other women receive combined oral contraceptives and antioxidant complex Selmevit.

The blood tests conduct on 19-21 days of the menstrual cycle before COC use (control group) or on 19-21 days of COC use after 1, 3, 6 and 12 cycles.

Also we investigate subjective tolerability, therapeutic effects, menstrual cycle control and adverse effects of COCs in women that have or have no antioxidant complex Selmevit

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-35 years
* Absence of contraindications for COC use
* Informed voluntary consent for examination

Exclusion Criteria:

* Age younger than 18 and older than 35 years
* Refusal or failure to comply with the study protocol
* Drug or alcohol dependence
* Psychiatric diseases
* Severe somatic and allergic diseases
* Pregnancy
* Malignancies
* Taking drugs that affect haemostasis, including hormonal contraceptives during 6 months before study beginning
* Cases of thrombosis among first-line relatives in family history
* Contraindications to the COC use under Eligibility Criteria of hormonal contraception (WHO, 2012)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-03 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Activated recalcification time | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in Activated partial thromboplastin time | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in Prothrombin time | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in International normalized ratio | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in D-dimer concentration | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in Fibrinogen concentration | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in Soluble fibrin-monomer complexes concentration | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in Platelet aggregation | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in Antithrombin III activity | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in Reserve plasminogen index | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in Erythrocyte Lipoperoxidation products, extractable in heptane and isopropanol | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in Malondialdehyde Concentration in Erythrocytes | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in Glutathion-S-transferase Activity in Erythrocytes | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Change from Baseline in Superoxide dismutase Activity in Erythrocytes | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)
Vitamin A and E plasma concentration | Baseline, 1, 3, 6 and 12 cycles of 4 weeks (between days 18 and 21 of each cycle)

SECONDARY OUTCOMES:
Frequency of adverse effects | 12 cycles of 4 weeks
Subjective tolerability of contraceptives | 12 cycles of 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tyumen State Medical Academy, Tyumen, Russia